CLINICAL TRIAL: NCT01618318
Title: Cross Sectional Study to Evaluate and Associate Clinical and Laboratory Features of People With Allergic and Non-allergic Asthma
Brief Title: Glasgow Asthma and Allergy Study
Acronym: GLAAS
Status: Completed | Type: Observational
Sponsor: National Services for Health Improvement Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 12/WS/0049
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Asthma; Allergy
Keywords: Asthma; Allergy; Diagnosis; Correlation study
MeSH Terms: conditions — Asthma; Hypersensitivity; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General asthma population: People with asthma, aged 18 years and over, non smoker, all severities of disease, regardless of treatment, broad inclusion and few exclusion criteria.

SUMMARY:
In the past, doctors separated people with asthma into two groups, those with "allergic asthma" (about 2/3rds of people) and those with "non-allergic asthma". These labels are not much used now as the treatments for all people with asthma don't depend on this classification. However, new treatments for asthma may become available and the classification may again become important. It could be useful for clinicians to know how to identify which patients are likely to benefit from particular treatments.

Additionally, some new blood tests are becoming available and some of these might help to categorise the type of asthma people have. What the study hopes to do is to identify patient features which make a diagnosis of "allergic asthma" more likely and to see which new blood tests are most likely to be helpful in confirming this diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years old and over with a diagnosis of asthma and having received at least two prescriptions for any asthma medication in the last 12 months, who have signed an informed consent form prior to initiation of any study-related procedure

Exclusion Criteria:

* under 18 years
* current smokers
* unwilling or unable to give informed consent
* a clinical diagnosis of COPD
* a history of anaphylaxis (skin prick test)
* participated in any clinical study in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with asthma, non smoker, aged 18 and over.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Serum periostin level | 1 day
  This is a cross sectional study. Participants will be assessed and tests conducted at a single visit

SECONDARY OUTCOMES:
skin prick test | 1 day
Serum total IgE | 1 day
Blood eosinophil count | 1 day
Blood neutrophil count | 1 day
Blood CD4 cells that are positive for CRTh2 | 1 day
Blood eosinophils expressing CRTh2 | 1 day
Spirometry | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: John A Haughney, MB ChB, Principal Investigator — NSHI Ltd
Locations (1):
- NSHI Ltd, Dartford, Kent, United Kingdom